CLINICAL TRIAL: NCT02574468
Title: Effect of Topical Dexamethasone on Histologic Response of Human Dental Pulp
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyed Amir Mousavi, Assistant professor of endodontics, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91_509
Record Dates: First submitted 2015-10-03; First posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Vital Pulp Therapy
Keywords: Dexamethasone; Direct pulp capping; MTA; pulpotomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DPC+Dexa (Active Comparator): forty intact premolars were randomly assigned to 1 of 4 treatment groups (n=10): I) DPC, II) MP, III) DPC+dexamethasone, and IV) MP+dexamethasone. After administration of local anesthesia (3% mepivacaine plain; Septodont, Cedex, France) dental rubber dam was applied and tooth surface disinfected with 2% chlorhexidine gluconate. Occlusal cavity was prepared using high speed diamond fissure bur and buccal pulp horn was mechanically exposed (approximately 1.2 mm in diameter) using a sterile high speed carbide round bur. In MP, depth of penetration to the pulp was 0.5 mm
  Interventions: Drug: Dexamethasone applied on pulp or Dexamethasone did not applied on pulp; Procedure: DPC or MP
- MP+Dexa (Active Comparator): forty intact premolars were randomly assigned to 1 of 4 treatment groups (n=10): I) DPC, II) MP, III) DPC+dexamethasone, and IV) MP+dexamethasone. After administration of local anesthesia (3% mepivacaine plain; Septodont, Cedex, France) dental rubber dam was applied and tooth surface disinfected with 2% chlorhexidine gluconate. Occlusal cavity was prepared using high speed diamond fissure bur and buccal pulp horn was mechanically exposed (approximately 1.2 mm in diameter) using a sterile high speed carbide round bur. In MP, depth of penetration to the pulp was 0.5 mm
  Interventions: Drug: Dexamethasone applied on pulp or Dexamethasone did not applied on pulp; Procedure: DPC or MP

INTERVENTIONS:
Drug: Dexamethasone applied on pulp or Dexamethasone did not applied on pulp — on half of cases we put dexamethasone on pulp on other half we did not put dexamethasone on pulp
Procedure: DPC or MP — on half of cases we treat teeth with DPC(Direct Pulp Cap) on other half we treat teeth with MP(Miniature Pulpotomy)

SUMMARY:
Abstract Aim The aim of this randomized clinical trial was to histologically investigate possible effects of dexamethasone application on pulp tissue healing during one step mineral trioxide aggregate (MTA)-direct pulp capping (DPC) and miniature pulpotomy (MP) in healthy human premolar teeth.

Methodology Forty intact premolar teeth of 10 orthodontic patients, scheduled for extraction, were randomized for DPC (n=20) or MP (n=20). A high speed bur under copious water coolant was used for mechanical exposing of buccal pulp horn site. Prior to sealing with white ProRoot MTA, 10 out of twenty pulpal wounds of each group were randomly received dexamethasone. Cavities were restored with glass ionomer. Teeth vitality was evaluated in 7, 21, 42, and 60 day follow-ups. Signs and/or symptoms of irreversible pulpitis or pulp necrosis were considered as failure. After 60 days, the teeth were extracted and submitted for histological examination. Kruskal-Wallis and Fisher exact tests were used for statistical analysis of the data (P=0.05).

HTTP://www.accessdata.fda.gov/scripts/cred/drugsatfda

DETAILED DESCRIPTION:
Clinical procedures All clinical procedures took place at private office of first author (J.G.). Using simple randomization procedures (computerized random numbers), forty intact premolars were randomly assigned to 1 of 4 treatment groups (n=10): I) DPC, II) MP, III) DPC+dexamethasone, and IV) MP+dexamethasone. After administration of local anesthesia (3% mepivacaine plain; Septodont, cedax, France) dental rubber dam was applied and tooth surface disinfected with 2% chlorhexidine gluconate. Occlusal cavity was prepared using high speed diamond fissure bur and buccal pulp horn was mechanically exposed (approximately 1.2 mm in diameter) using a sterile high speed carbide round bur. In MP, depth of penetration to the pulp was 0.5 mm. All of the cavity preparation procedures were intermittently performed under copious water coolant and light hand pressure. Using a sterile 5.25% NaOCl-soaked cotton pellet, bleeding from the exposure site was controlled and 2ml of sterile saline rinsed off NaOCl residues. For blinding the practitioner to the materials, dexamethasone (Dr.abidi, Tehran, Iran) and placebo were held in identical light proof syringes and numbered for each tooth according to the randomization schedule. Each tooth was assigned an order number and its pulpal wound received the solution in the corresponding prepacked syringe prior to sealing off the exposure site with white ProRoot MTA (Dentsply, Tulsa, OK); MTA was mixed according to the manufacturer's directions and a wet cotton pellet was placed over the material for 10 minutes. Eventually, the coronal cavity was restored with light cure resin modified glass ionomer (Fuji II LC; GC Corporation, Tokyo, Japan) and cured for 40 seconds using a curing light. All clinical procedures were performed by the same practitioner (J.G.). All patients took 400 mg of ibuprofen (as a single dose) for postoperative pain control. Pulp and periapical status were clinically (7, 21, 42, and 60 days) and radiographically evaluated (42, and 60 days) during the study. Clinical and radiographic signs and/or symptoms of irreversible pulpitis or pulp necrosis were considered as treatment failure. On the 60th day teeth were extracted atraumatically and prepared for submission to the oral pathology department for processing.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult patients who had four intact fully developed upper and lower premolars needed to be extracted because of his/her orthodontic treatment plan were eligible

Exclusion Criteria:

* Exclusion criteria were history of previous trauma
* clinical and/or radiographic caries
* restorations, periodontal problems
* intake of anti-inflammatory medication before (over the last couple of weeks) and during the study
* known allergy and/or contraindications to dexamethasone

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Histologic Evaluation of pulp for inflammation | one year
  measure number of inflammatory cells for amount of inflammation
Histologic Evaluation of pulp for calcified bridge | one year
  measure thickness of calcified bridge on the pulp
Histologic Evaluation of pulp for odontoblast layer | one year
  measure odontoblastic cells on odontoblast layer